CLINICAL TRIAL: NCT01897675
Title: Is Loop Drainage of a Cutaneous Abscess in the Emergency Department as Effective as Incision and Drainage With Packing?
Brief Title: A Comparison of Techniques for Treating Skin Abscesses
Acronym: LoopDrainage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Elissa Schechter-Perkins, Assistant Professor of Emergency Medicine, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-32294
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Cutaneous Abscess
Keywords: Cutaneous Abscess; Emergency Department
MeSH Terms: conditions — Emergencies | interventions — Drainage; Drug Packaging; Drug Implants

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incision and Drainage with Packing (Active Comparator): Abscess is cared for in the standard fashion, using an incision and drainage with packing (wick) placement. Packing to be changed every 2-3 days, at the discretion of the treating clinician, until abscess is considered resolved
  Interventions: Procedure: Incision and Drainage with packing (wick) placement
- Loop Drainage (Experimental): Abscess is cared for using a minimally invasive abscess drainage with loop placement technique. Two (or more) stab incisions are made in the abscess, the cavity is probed and pus is drained, and a vessel loop is inserted and tied off. The patient manipulates the loop 3 times per day, and removes the loop when all redness is gone and no more pus is present
  Interventions: Procedure: Abscess drainage with loop placement

INTERVENTIONS:
Procedure: Incision and Drainage with packing (wick) placement
  Arms: Incision and Drainage with Packing
Procedure: Abscess drainage with loop placement
  Arms: Loop Drainage

SUMMARY:
Management of abscesses traditionally involves incision and drainage (I&D). Abscesses are frequently are "packed" or stented open with the presence of a wick, and traditional care requires re-visits every 2-3 days to have the packing removed and replaced, until finally the abscess cavity has closed, usually 1-2 weeks after initial presentation.

Recently there have been attempts to employ less invasive techniques for abscess management. One novel technique, "loop drainage", has been reported in case reports/case series for management of a variety of types of abscesses in the surgical subspecialty literature.

We propose to conduct a randomized prospective study comparing the efficacy of the loop drainage technique with the traditional incision and drainage technique of abscess management.

Patients presenting to the main or urgent care areas of the Emergency Department at Boston Medical Center for treatment of an abscess will be considered for enrollment as potential subjects. After the treating clinician identifies the patient as an appropriate subject, a Research Associate (RA) will approach the patient and obtain written informed consent to enroll in the study. The subject will then be randomized to the management arm of either loop drainage or traditional I&D. The clinician will fill out a data sheet describing the abscess characteristics, and then perform either loop drainage or incision and drainage, depending on randomization and the subject will fill out a satisfaction survey. Fourteen days after initial visit, subjects will return for follow-up. The subject will fill out a satisfaction survey, and a study investigator blinded to the treatment group will assess the subject for abscess resolution, cosmetic outcome, number of follow-up visits, and complications.

The study investigators will then compare outcomes between the two study groups.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient over 18 years of age
* Presenting to the Boston Medical Center main Emergency Department or Urgent Care area for initial treatment of a skin abscess
* English speaking
* Able to provide written informed consent
* Willing to return in 14 days for follow-up visit
* Able to give a telephone number for follow-up contact

Exclusion Criteria:

* Previously treated for this abscess
* Altered mental status
* Patients with active psychiatric issues that preclude their ability to provide informed consent
* Previously enrolled in the study
* Abscess is not amenable to treatment by an Emergency Physician in the Emergency Department
* Abscess is post-operative or post-procedure
* Clinician determines abscess is not amenable to drainage by particular method
* Abscess is too small for packing or loop
* Need for hospital admission

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03-09 (Actual)

PRIMARY OUTCOMES:
Abscess Resolution | 14 days
  If no, which sign is present (check all that apply):
  1. Fluctuance
  2. Drainage
  3. Induration
  4. Warmth
  5. Tenderness
  6. Other __________

SECONDARY OUTCOMES:
Patient Satisfaction Immediately After Procedure | Time 0
  How Satisfied is Patient Immediately after Procedure (likert scale) Did Patient Feel Discomfort During Procedure (likert scale)
Cosmetic Outcome | 14 days
  Appearance according to wound scale
  Wound Scale (presence or absence of)
  1. Step-off of borders
  2. Contour irregularities
  3. Wound margin separation
  4. Edge inversion
  5. Excessive distortion
  6. Overall appearance
Patient Satisfaction after Abscess Resolution | 14 Days
  Patient Satisfaction with:
  Number of Follow Up Visits (likert scale) Cosmetic Appearance (likert scale) Pain (likert scale) Overall abscess care (likert scale
Number of Follow Up Visits | 14 days
  Number of follow-up visits made to either Emergency Department or outpatient clinic for abscess care
Number of Complications | 14 days
  need for new incision in the same abscess, extension of the original incision, starting antibiotics, changing antibiotics, admission

CONTACTS AND LOCATIONS:
Overall Officials: Elissa Schechter-Perkins, MD, MPH, Principal Investigator — Boston Medical Center
Locations (1):
- Boston University Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McNamara WF, Hartin CW Jr, Escobar MA, Yamout SZ, Lau ST, Lee YH. An alternative to open incision and drainage for community-acquired soft tissue abscesses in children. J Pediatr Surg. 2011 Mar;46(3):502-6. doi: 10.1016/j.jpedsurg.2010.08.019. PMID 21376200
- [Background] Ladd AP, Levy MS, Quilty J. Minimally invasive technique in treatment of complex, subcutaneous abscesses in children. J Pediatr Surg. 2010 Jul;45(7):1562-6. doi: 10.1016/j.jpedsurg.2010.03.025. PMID 20638546
- See also: Video of Loop Drainage Technique for Abscess care — http://vimeo.com/19580472